CLINICAL TRIAL: NCT06297031
Title: The Effect of Heat Application to the Sacral Region During The First Stage of Labor On the Pain Level and the Obstetric Outcomes
Brief Title: Heat Application to the Sacral Region and Pain Level During the First Stage of Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Demiroglu Bilim University (Other)
Responsible Party: Principal Investigator, Tulay Kavlak, Assistant Professor, Istanbul Demiroglu Bilim University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020/20
Record Dates: First submitted 2024-02-21; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Heat Exposure; Labor Pain; Apgar Score; Duration of Labor
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- heat application (Experimental): women in the intervention group were treated with hot water application to the sacral region during the first stage of labor. When the cervical dilatation was 3-4 cm, 5-6 cm and 7-8 cm, heat application was applied a total of 3 times.
  Interventions: Other: heat application
- no heat application (No Intervention): No treatment was performed on women in the control group during the study. In the clinic, women's cervical dilatation is routinely checked by the midwife every 2-3 hours, and the progress of labor is monitored by fetal heart rate and fetal monitoring

INTERVENTIONS:
Other: heat application — • Thermophore Application: Before the application, the thermophore was wrapped in a towel to prevent skin damage. Studies in the literature indicate that the surface temperature of the thermophore should be 38-45 °C. For this reason, water with a temperature of 70°C when measured with a thermometer was added into the thermophore. Similarly, studies in the literature indicate that thermophore application should be applied for 10-30 minutes. Therefore, the application takes 20 minutes. The researcher stayed with the woman for 20 minutes.
  Arms: heat application

SUMMARY:
The aim of this study was to determine the effect of hot application applied to the sacral region during first stage of labor on women's pain level and labor process.

DETAILED DESCRIPTION:
It is stated that the pain experienced during labor, which is a physiological process, creates stress and anxiety in women and increases the risk of maternal and neonatal complications. Therefore, keeping labor pain under control is important from an obstetrical perspective. Pain experienced during labor is caused by dilatation of the cervix and uterine contractions, and occurs in different regions at each stage of labor. Due to the descent of the fetal head into the pelvis and the pressure it puts on the lumbosacral plexus, the mother feels pain in her back, waist, legs and hips, especially in the first stage of labor. Although pharmacological and non-pharmacological methods are used in the management of labor pain, they have disadvantages such as experiencing drug-related side effects due to pharmacological methods, causing undesirable effects in the woman and the fetus, the woman not being able to actively participate in the labor and not being able to remember what happened during labor.

ELIGIBILITY:
Inclusion Criteria:

* Women were over 18 years of age
* Primipara
* Volunteered to participate in the study
* Were in the latent phase of labor (cervical dilatation 1-2 cm)
* Had a single fetus in vertex presentation
* Had no history of pregnancy complications
* Had not undergone any intervention in the sacral region were included in the study

Exclusion Criteria:

* Applied pharmacological pain control methods in the first stage of labor
* Had a cesarean section decision at any stage

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 134 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Change From Baseline labor Pain at three times | The pain was evaluated three times during labor
  It will be assessed three times during the first stage of the labor with Number Rating Scale. Pain intensity measured on a Number Rating Scale with scores ranging from 0 - 10. Pain increases as the score increases. The high point describes bad outcome.

SECONDARY OUTCOMES:
Duration of the first stage of labor | through study completion, an average of 1 day
  The time between the start of the pain expressed by the woman and the moment she was taken to the delivery table was calculated by the researcher and called the first stage of labor. The researcher used clock to calculate the duration
Change From Baseline APGAR score after delivery | After delivery in two times at first and fifth minutes through study completion, an average of 1 day
  The scale is designed to determine the need for urgent intervention by assessing the condition of the newborn in order to reduce neonatal morbidity and mortality rates. A score of 0 represents the lowest level of functionality, while a score of 10 indicates optimal health. A score below 4 indicates that the newborn has significant respiratory distress that requires urgent medical attention
Change From Baseline Fetal Heart Rate | A total of three measurement results were obtained (after the cervical dilatation was evaluated as 3-4 cm, 5-6 cm and 7-8 cm)
  after the cervical dilatation Fetal Heart Rate was evaluated with monitor. the recommended level is 100 to 160 heart beat/minute

CONTACTS AND LOCATIONS:
Overall Officials: Tülay KAVLAK, Principal Investigator — Istanbul Demiroglu Bilim University
Locations (1):
- Demiroglu Bilim University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goswami S, Jelly P, Sharma SK, Negi R, Sharma R. The effect of heat therapy on pain intensity, duration of labor during first stage among primiparous women and Apgar scores: A systematic review and meta-analysis. Eur J Midwifery. 2022 Nov 28;6:66. doi: 10.18332/ejm/156487. eCollection 2022. PMID 36474673
- [Background] Kaur J, Sheoran P, Kaur S, Sarin J. Effectiveness of Warm Compression on Lumbo-Sacral Region in Terms of Labour Pain Intensity and Labour Outcomes among Nulliparous: an Interventional Study. J Caring Sci. 2020 Mar 1;9(1):9-12. doi: 10.34172/jcs.2020.002. eCollection 2020 Mar. PMID 32296653